CLINICAL TRIAL: NCT00055575
Title: Cholinergic Modulation of Cognition and Emotion in Mood Disorders: Functional Neuroimaging Studies
Brief Title: Cholinergic Modulation of Condition and Emotion in Mood Disorders: Functional Neuroimaging Studies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 030108; 03-M-0108
Record Dates: First submitted 2003-03-06; First posted 2003-03-06 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2015-02-02

CONDITIONS: Mood Disorders; Healthy; Unipolar Depression; Bipolar Depression
Keywords: Scopolamine; Depression; fMRI; Cognition; Emotion; Brain; Bipolar Disorder; Major Depressive Disorder; MDD; Healthy Volunteer; HV
MeSH Terms: conditions — Mood Disorders; Depressive Disorder; Bipolar Disorder; Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Depressed Patients with Major Depression DIsorder (Experimental)
  Interventions: Drug: Scopolamine Nasal Spray
- Depressed Patients with Bipolar Disorder (Experimental)
  Interventions: Drug: Scopolamine Nasal Spray
- Healthy Control (Experimental)
  Interventions: Drug: Scopolamine Nasal Spray

INTERVENTIONS:
Drug: Scopolamine Nasal Spray

SUMMARY:
This study looks at the role of a specific brain chemical system in the mood and attention symptoms seen in major depression and bipolar disorders using functional brain imaging.

DETAILED DESCRIPTION:
1. Objective

   The goal of this research project is to evaluate the role of the cholinergic system in behavioral and cognitive symptoms observed in mood disorders in humans, using functional brain neuroimaging techniques. Specific aspects of behavior and cognition are impaired in mood disorders, including selective attention, set-shifting and memory; and there is also evidence that depressed subjects exhibit a mood congruent processing bias whereby they more readily process negatively toned information as compared to positively toned information. This cognitive pattern lends itself to evaluation with functional brain imaging, both in terms of identifying the anatomical correlates of the specific behavioral and cognitive deficits as well as characterizing the effects of pharmacological manipulation.

   Attention and memory functions are closely tied to the cholinergic neurotransmitter system. The cholinergic system is one of the neurotransmitter systems implicated in the pathophysiology of mood disorders. Evidence suggests that during major depressive episodes, the cholinergic system is hypersensitive to acetylcholine. Agents that enhance muscarinic cholinergic receptor function increase depressive symptoms in depressed subjects, and can produce symptoms of depression in healthy subjects. The preclinical literature more specifically implicates the muscarinic receptors and indicates that the use of muscarinic antagonists, in the context of animal models of depression, results in improvement in the behavioral analogs of depression.
2. Study Population

   The accrual ceiling for this protocol is 388 participants. 143 currently depressed patients with major depressive disorder, 100 currently depressed patients with bipolar disorder, and 145 healthy controls will participate in this study.
3. Design

   The antimuscarinic agent, scopolamine, will be administered in a double-blind, placebo controlled manner across all studies. Clinical ratings, cognitive tasks and neuroimaging will be conducted at various timepoints to evaluate the clinical effects of scopolamine on depression, to assess the acute mood response to scopolamine; and to study the neurobiological correlates of the clinical and behavioral drug effects.
4. Outcome Measures

The proposed inpatient or outpatient project investigates the role of cholinergic neurotransmission in the behavioral and cognitive symptoms observed in the depressed phase of both major depressive disorder (MDD) and bipolar disorder (BD). The studies proposed here will identify anatomical correlates of the mood congruent processing bias, working memory, attention and set-shifting deficits observed in depressed subjects. Further, these studies will evaluate the effects of the cholinergic antagonist, scopolamine, both on the performance deficits and on neural activity in brain regions recruited as subjects perform these tasks.

Dose escalation studies will be conducted to determine if higher doses of scopolamine will increase the antidepressant response rate in patients with major depressive disorder. Based on earlier work showing the predictive value in baseline neuroimaging data to predict treatment outcome, we will stratify participants at baseline into groups based on expected response to scopolamine treatment.

This approach is expected to reveal how neuromodulators influence processing in brain structures recruited to perform these tasks, both in healthy subjects and in major depressive disorders. The combined use of functional brain imaging and pharmacological manipulation to evaluate the role of neurotransmitter dysfunction in depression may direct us to potential therapeutic approaches.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with Major Depressive Disorder (MDD):

* Age 18-55
* Current diagnosis of MDD, as defined by DSM-IV criteria for recurrent MDD
* Current depressive episode
* Current IDS score in the moderately-to-severely depressed range
* Right handed
* Able to provide informed consent

Patients with Bipolar Disorder (BD):

* Age 18-55
* Current diagnosis of bipolar disorder, as defined by DSM-IV
* Current depressive episode
* Current IDS score in the moderately-to-severely depressed range
* Right handed
* Able to provide informed consent

Healthy Controls:

* Age 18-55
* Able to provide informed consent
* Medically healthy

EXCLUSION CRITERIA:

Patients MDD & BD:

* Serious suicidal ideation or behavior (with a current plan or intent), or current delusions or hallucinations
* Medical or neurological illnesses likely to affect physiology or anatomy
* History of drug or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM IV criteria)
* Current or past history of other axis I disorders that preceded the onset of MDD or BD
* Current pregnancy (documented by pregnancy testing within 24 hours prior to pilot studies and 24 hours prior to scanning)
* Current breast feeding
* General MRI exclusion criteria (including the presence of pacemakers, cochlear implants, surgical clips or metal fragments in their eyes or body parts)
* Vision and/or hearing problems severe enough to interfere with testing
* Electrocardiographic evidence of ischemia, arrhythmia, conduction defect, or myocardial infarction
* Current blood pressure of >140 mm Hg or < 90 mm Hg systolic, or > 90 mm Hg diastolic (due to the potential cardiovascular effects of scopolamine and physostigmine)
* Clinically significant cerebrovascular or cardiovascular disease, hypertension, congestive heart disease, angina pectoris, advanced arteriosclerosis, gross neurological impairment, hyperthyroidism, known hypersensitivity or idiosyncrasy to anticholinergic agents, glaucoma, renal or hepatic impairment
* Clinical history of glaucoma or narrow angle glaucoma (due to the possibility of exacerbation of this condition by scopolamine)
* Age of onset greater than 45 years (to reduce the biological heterogeneity encompassed by the MDD and BD criteria, since subjects with a late age-at onset for depression have a far greater likelihood of having MRI correlates of cerebrovascular disease than age-matched, healthy controls or age-matched, early-onset depressives)
* Exposure within two weeks to medications likely to effect cerebral blood flow and metabolism or likely to interact with anti-cholinergic medications (e.g. narcotics or anti-cholinergic agents)- as verified by history and urine drug screen
* HIV positive status
* Weight over 275 pounds

Healthy Controls:

* Medical or neurological illness
* Current pregnancy (documented by pregnancy testing within 24 hours prior to pilot studies and 24 hours prior to scanning)
* Current breast feeding
* General MRI exclusion criteria (including the presence of pacemakers, cochlear implants, surgical clips or metal fragments in their eyes or body parts)
* Vision and/or hearing problems severe enough to interfere with testing
* Electrocardiographic evidence of ischemia, arrhythmia, conduction defect, or myocardial infarction
* Current blood pressure of >140 mm Hg or < 90 mm Hg systolic, or > 90 mm Hg diastolic (due to the potential cardiovascular effects of scopolamine and physostigmine)
* Clinically significant cerebrovascular or cardiovascular disease, hypertension, congestive heart disease, angina pectoris, advanced arteriosclerosis, gross neurological impairment, hyperthyroidism, known hypersensitivity or idiosyncrasy to anticholinergic agents, glaucoma, renal or hepatic impairment
* Clinical history of glaucoma or narrow angle glaucoma (due to the possibility of exacerbation of this condition by scopolamine)
* HIV positive status
* Weight over 275 pounds

For BD patients being recruited for the scopolamine efficacy trial, they may forgo imaging and thus will not be excluded for imaging related exclusion criteria (including general MRI exclusion criteria and vision and/or hearing problems).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2003-02-27; Primary Completion 2015-02-02 (Actual); Study Completion 2015-02-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the antidepressant effects of the antimuscarinic agent scopolamine | 5 to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Elliott R, Rubinsztein JS, Sahakian BJ, Dolan RJ. Selective attention to emotional stimuli in a verbal go/no-go task: an fMRI study. Neuroreport. 2000 Jun 5;11(8):1739-44. doi: 10.1097/00001756-200006050-00028. PMID 10852235
- [Background] Murphy FC, Sahakian BJ, Rubinsztein JS, Michael A, Rogers RD, Robbins TW, Paykel ES. Emotional bias and inhibitory control processes in mania and depression. Psychol Med. 1999 Nov;29(6):1307-21. doi: 10.1017/s0033291799001233. PMID 10616937
- [Background] Murray LA, Whitehouse WG, Alloy LB. Mood congruence and depressive deficits in memory: a forced-recall analysis. Memory. 1999 Mar;7(2):175-96. doi: 10.1080/741944068. PMID 10645378
- [Derived] Furey ML, Drevets WC, Hoffman EM, Frankel E, Speer AM, Zarate CA Jr. Potential of pretreatment neural activity in the visual cortex during emotional processing to predict treatment response to scopolamine in major depressive disorder. JAMA Psychiatry. 2013 Mar;70(3):280-90. doi: 10.1001/2013.jamapsychiatry.60. PMID 23364679